CLINICAL TRIAL: NCT06775574
Title: Prognostic Significance of the Lung Immune Prognostic Index (LIPI) in Postoperative Clear Cell Renal Cell Carcinoma: a Multicenter Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 0361-01
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: ccRCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients with dNLR < 3 and LDH levels below the upper limit of normal
- Cohort 2: Patients with dNLR ≥ 3 and LDH levels above the upper limit of normal

SUMMARY:
This retrospective study included 704 patients with ccRCC who underwent radical or partial nephrectomy. Patients were stratified into the LIPI good group and the intermediate/poor (int./poor) group based on dNLR (≥ 3) and LDH (≥ 245 U/L) levels. Propensity score matching (PSM) was used to adjust for baseline differences and minimize selection bias. Kaplan-Meier survival curves and Cox regression models were employed to evaluate the impact of LIPI and other clinical factors on recurrence-free survival (RFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed with ccRCC;
2. Underwent radical or partial nephrectomy.

Exclusion Criteria:

1. presence of concurrent malignancies;
2. missing data or failure to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study included 704 patients with ccRCC who underwent radical or partial nephrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 704 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | 5 years
recurrence-free survival (RFS) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China